CLINICAL TRIAL: NCT05666232
Title: Renal Resistive Index and Myocardial Performance Index for Early Prediction of Acute Kidney Injury After Living Donor Liver Transplantation
Brief Title: Renal and Cardiac Risk Factors of AKI After Liver Transplantation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Other Study IDs: MD.22.09.699
Record Dates: First submitted 2022-12-18; First posted 2022-12-27 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Acute Kidney Injury; Acute Renal Injury; Liver Transplant; Complications
Keywords: 2-D Echocardiography; Two-Dimensional Echocardiography; renal resistive index; myocardial performance index; diagnostie test accuracy; sensitivity and specificity
MeSH Terms: conditions — Acute Kidney Injury; Hypersensitivity | interventions — Echocardiography; Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: renal resistive index and myocardial performance index — Transthoracic echocardiography and transabdominal ultrasonography will be performed before induction of anesthesia, after termination of operation and before transmission to ICU and then daily for the early seven postoperative days.
  RRI = (peak systolic velocity - end diastolic velocity) ∕ peak systolic velocity: Then, we will obtain the mean RRI from the above three measurements.
  We will consider RRI ≥0.7 as abnormal and define it as subclinical AKI.
  Myocardial performance index (using tissue doppler) =
  (isovolumetric contraction time + isovolumetric relaxation time) / ejection time. We will consider MPI ≥0.4 as abnormal and define it as subclinical LV dysfunction.
  Other Names: echocardiography; ultrasonography

SUMMARY:
Background: Liver transplantation (LT) is an extensive operation with various factors contributing to the development of acute kidney injury in the perioperative period. Early diagnosis of AKI can improve clinical outcomes in LT recipients. Renal resistive index is measured in renal arteries and high resistive values are associated with more adverse cardiovascular events and renal failure progression. Myocardial performance index reflects overall cardiac function rather than systolic or diastolic function alone.

Aim of the study: to investigate whether combined doppler renal resistive index and myocardial performance index could predict early postoperative acute kidney injury in living donor liver transplant recipients.

Study design: a prospective observational study that will be conducted at Liver Transplantation Unit at Mansoura University on 105 consecutive living donor liver transplant recipients.

Methods: Renal resistive index (assessed by transabdominal ultrasound) and myocardial performance index (assessed by transthoracic echocardiography) will be measured just before operation, on termination of operation and then daily in the intensive care unit for 7 days. Patients will be observed for development of acute kidney injury.

DETAILED DESCRIPTION:
This study aims to investigate whether combined doppler renal resistive index (RRI) assessed by transabdominal sonography and myocardial performance index (MPI) assessed by transthoracic echocardiography could predict early postoperative acute kidney injury in living donor liver transplant recipients.

The primary outcome is the predictive value of renal resistive index and myocardial performance index for the onset of early post living donor liver transplant acute kidney injury.

This prospective observational study will be conducted at Liver Transplantation Unit at Mansoura University from November 2022 till fulfillment of sample size after obtaining approval from Institutional Review Board (IRB). One hundred and five consecutive LDLT recipients will participate in this study after obtaining informed consents. They will be observed for the development of early postoperative acute kidney injury.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing right-lobe living-donor liver transplantation

Exclusion Criteria:

* preoperative renal impairment (GFR < 60 ml/min/1.73 m2)
* known renal artery stenosis
* patient who underwent previous nephrectomy
* ischemic heart disease (patient who takes anti-ischemic measures as prescribed by a consultant cardiologist)
* Patient with arrthymia or who develop persistent intraoperative arrythmia

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing living donor liver transplantation at gastrointestinal surgery center at Mansoura University - Mansoura, Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
early acute kidney injury (AKI) | in the early 48 postoperative hours
  international Club of Ascites' revised classification of AKI in cirrhotic patients as a 0.3 mg/kg increase in serum creatinine

SECONDARY OUTCOMES:
stage of AKI | in the early 48 postoperative hours
  Stage (1): serum creatinine increase 1.5- 1.9 times base line; or serum creatinine increase more than 0.3mg/dl. Stage (2): serum creat. Increase 2-2.9 times baseline. Stage (3): serum creat. Increase 3 times baseline ; or s.creat increase to 4mg/dl; or initiation of renal replacement therapy.
late AKI | within 7 days
  International Club of Ascites' revised classification of AKI in cirrhotic patients as a 0.3 mg/kg increase in serum creatinine or >= 50% increase in the basal serum creatinine
length of ICU stay | 3 months after transplant
  duration of ICU stay (days) in survived patients
length of hospital stay | 3 months after transplant
  duration of ICU stay (days) in survived patients
three-month mortality | 3 months after transplantation
  all-cause mortality
delayed renal function | 3 months after transplantation
  serum creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Amr Yassen, MD, Study Chair — Mansoura University Hospital

IPD SHARING:
Plan to Share IPD: Yes
The anonymized patient data will be available on reasonable request after approval of the local IRB.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: within 3 months